CLINICAL TRIAL: NCT01954680
Title: COGFLEX: Pilot Translational Intervention of Pediatric Bipolar Disorder
Brief Title: Retrain Your Brain in Children/Adolescents With Bipolar Disorder: A Pilot Study
Acronym: COGFLEX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bradley Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0195-07 COGFLEX; R21MH096850 (NIH); R33MH096850 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-10-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder; Pediatric Bipolar Disorder; Childhood-onset Bipolar Disorder
Keywords: bipolar disorder; child; adolescent
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: R21 phase was an open phase 1a trial for feasibility and acceptability with enrollment goal including intervention development of 20.
  R33 phase enrollment goal of 40 including double-blind placebo-controlled randomized trial of 2 versions of video game potential intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Neither participant nor independent evaluator knows group assignment in R33 phase randomized controlled trial.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COGFLEX-skill building levels (Experimental): In the R33, children will be randomized to receive either COGFLEX with skill-building levels or just baseline/non-probabilistic trials. All children will play COGFLEX twice per week for 8-weeks.
  Interventions: Behavioral: COGFLEX-skill building levels
- COGFLEX-control condition (Experimental): In the R33, children will be randomized to receive either COGFLEX with skill-building levels or the control condition--which is just baseline/non-probabilistic trials. All children will play COGFLEX twice per week for 8-weeks.
  Interventions: Behavioral: COGFLEX-control condition

INTERVENTIONS:
Behavioral: COGFLEX-skill building levels — COGFLEX--in English-- is a computer game designed to build up a specific skill that our work has shown is impaired in children and adolescents with bipolar disorder).
  In the R33, children will be randomized to receive either COGFLEX with skill-building levels or COGFLEX-control condition which is just baseline/non-probabilistic trials.
  All children will play COGFLEX twice per week for 8-weeks.
  This same approach has shown great success in many psychiatric disorders including schizophrenia.
  This is the first such study in children/adolescents with bipolar disorder.
  Other Names: COGFLEX is a computer assisted cognitive remediation
  Arms: COGFLEX-skill building levels
Behavioral: COGFLEX-control condition — In the R33, the control condition will be the same COGFLEX "game"--but just baseline/non-probabilistic trials. All children will play COGFLEX twice per week for 8-weeks.
  Arms: COGFLEX-control condition

SUMMARY:
The main aim of this study is to test a new, non-medication computer-based potential treatment for bipolar disorder in children and adolescents.

In the study, children and adolescents with bipolar disorder will come to our lab at Bradley Hospital 2-times per week for 8-weeks to "play" a custom computer "game" designed to retrain the brain--to build a skill that my work has shown is impaired in children/adolescents with bipolar disorder.

Before and after this 8-week trial, children will have a special magnetic resonance imaging (MRI) scan.

This is a test of feasibility--meaning we want to see if the 8-week trial results in brain changes.

If it does, we will conduct a second study to see if it improves how bipolar children function--i.e., if it helps their illness.

DETAILED DESCRIPTION:
Prior studies have shown that "computer assisted cognitive remediation"--meaning using computer "games" to build up a skill that has been shown to be impaired in a specific disorder--can result in improvement in psychiatric illnesses--including schizophrenia.

This will be the first National Institute of Mental Health (NIMH)-funded study to use this "retrain your brain" approach in children and adolescents with bipolar disorder.

During this study, we are seeking 40 children and adolescents with bipolar disorder to:

* come to our lab at Bradley Hospital in East Providence R.I. twice per week (each lasting 1 hour) to "play" a special computer game for a total of 8 weeks
* to have a special MRI before and after this 8-week trial to see if our "game" improves brain activity
* it does NOT matter if your child is already on medications--they can continue during this study
* all children/adolescents with bipolar disorder are welcome--as long as they do NOT have implanted metal (no braces, no cochlear implants, etc) because of magnetic resonance imaging (MRI) safety.

This is a test of feasibility--meaning we want to see if the 8-week trial results in brain changes.

If it does, we will conduct a second study to see if it improves how bipolar children function--i.e., if it helps their illness.

ELIGIBILITY:
Inclusion Criteria:

* 7-17 years old
* bipolar disorder type I preferred (at least 1 week of mania)

Exclusion Criteria:

* no implanted metal (no braces, no cochlear implants)
* can not have full Diagnostic and Statistical Manual 4th Edition (DSM-IV) autistic disorder
* no active drug/alcohol abuse/dependence

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in functional magnetic resonance imaging (fMRI) brain activation | Change from week 1 to week 8
  We will compare functional magnetic resonance imaging (fMRI) brain activation from week 1 (before intervention starts) to week 8 (after intervention is complete).

SECONDARY OUTCOMES:
Change in Clinician global Impression Improvement-Irritability | Change from week 1 to week 8
  Clinician global Impression Improvement-Irritability

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickstein, M.D., Principal Investigator — Bradley Hospital/Alpert Medical School of Brown University
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States